CLINICAL TRIAL: NCT03484390
Title: Effects of Mindfulness on PTSD: A Community-Based Clinical Trial Among Trauma Survivors
Brief Title: Effects of Mindfulness on PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Autumn Gallegos, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 64139
Record Dates: First submitted 2018-03-22; First posted 2018-03-30 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Mindfulness; Stress Disorder, Posttraumatic
Keywords: mindfulness; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction (Experimental): The MBSR program is a manualized course that includes meditation, relaxing movement, and breathing. A certified MBSR instructor will teach the courses in a group-based format for 120 minute sessions, once per week for eight weeks.
  Interventions: Behavioral: Mindfulness-based stress reduction
- Wellness Group (Active Comparator): The Wellness control group uses a health education manual that provides information on various aspects of health, including diet, physical activity, sleep, stress management, and communication. The manual is used during weekly check-in phone calls for an 8-week period.
  Interventions: Behavioral: Wellness Group

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction
  Arms: Mindfulness-based stress reduction
Behavioral: Wellness Group
  Arms: Wellness Group

SUMMARY:
The purpose of this randomized control trial is to examine the effects of a Mindfulness-Based Stress Reduction (MBSR) program on women with posttraumatic stress disorder related to intimate partner violence.

DETAILED DESCRIPTION:
Posttraumatic stress disorder is a prevalent, chronic, and debilitating disorder characterized by a reduced capacity to adapt to stressors, marked by poor regulation in the following domains: emotion, attentional function, and physiological stress. Mindfulness-based stress reduction (MBSR) holds promise for treating symptoms of trauma and PTSD as evidence suggests it targets these domains. The central hypothesis is that MBSR, which teaches non-judgmental awareness, can improve emotion regulation and attentional function, and diminish physiological stress dysregulation, which in turn will improve PTSD symptoms. We will examine changes in stress capacity and PTSD symptom severity among women survivors of intimate partner violence with PTSD after participation in an MBSR program.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Women
* 18-64 years of age
* Victim of IPV
* Meet diagnostic criteria for PTSD
* No or stable use of medications (including, for example, beta blockers).

Exclusion Criteria:

* There is suspicion or evidence of dementia or cognitive impairment (Mini-Mental State Examination score < 24) or inability to provide informed consent
* They have ever been a perpetrator of IPV
* History of schizophrenia or bipolar I disorder; current suicidality with either plan, intent, or a suicide attempt in the past 6 months
* Active substance dependence or in remission < 3 months
* Cardiovascular conditions (e.g., congestive heart failure, pacemaker, prior myocardial infarction)
* The age range was chosen to reduce heterogeneity in this pilot study, as aging is associated with changes in emotion regulation, attention, and PNS tone.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms Checklist (PCL-5) | 12 weeks
  The PTSD Symptoms Checklist (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 asks respondents to rate how much they have been bothered by particular PTSD symptoms in the past month on a 0-4 scale.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | 12 weeks
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report measure that assesses emotion dysregulation in six domains: nonacceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
Heart rate variability | 12 weeks
  To assess cardiovascular measures, ECG, basal thoracic impedance (Z0), the first derivative of the impedance signal (dZ/dt), and continuous strain gauge signal, will be obtained (BioNex Mainframe, Mindware Technologies, Gahanna, OH). Three disposable ECG electrodes will be placed in a lead II configuration to record the ECG signal. Four additional disposable patient ECG spot electrodes (2 current and 2 recording electrodes) will be used to obtain the Z0 and dZ/dt signals. A strain gauge will be secured around the lower chest to record respiration rate. The BioNex will be connected to a laptop: signals will be conditioned and collected (1000 Hz sampling; 5 Hz for strain gauge) through an integrated A/D board, and written to disk and later scored (with Mindware software).
Useful Field of View Test (UFOV) | 12 weeks
  The Useful Field of View Test (UFOV) is a computerized test with 3 assessments: speed of processing; selective attention; divided attention. The test determines the minimum display duration at which participants can process information for increasingly difficult subtests and is the primary outcome for prior studies of speed of processing training.
Five-Facet Mindfulness Questionnaire (FFMQ) | 12 weeks
  The Five-Facet Mindfulness Questionnaire assesses five factors that represent mindfulness as it is currently conceptualized: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn Gallegos, PhD, Principal Investigator — University of Rochester
Locations (1):
- Monroe County Family Court, Rochester, New York, United States

REFERENCES:
- [Derived] Gallegos AM, Heffner KL, Cerulli C, Luck P, McGuinness S, Pigeon WR. Effects of mindfulness training on posttraumatic stress symptoms from a community-based pilot clinical trial among survivors of intimate partner violence. Psychol Trauma. 2020 Nov;12(8):859-868. doi: 10.1037/tra0000975. Epub 2020 Sep 24. PMID 32969703